CLINICAL TRIAL: NCT05325879
Title: Investigation of the Relationship of Cervical Region Tension With Vagal Function and Gastrointestinal Symptoms
Brief Title: Relationship of Cervical Region Tension With Vagal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Yasemin Özel Aslıyüce, Research Assistant, Hacettepe University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: HUSpine014
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Gastrointestinal Diseases; Autonomic Nervous System Disease
Keywords: vagus nerve; muscle tonus; Autonomic Nervous System Diseases; Pain Threshold
MeSH Terms: conditions — Gastrointestinal Diseases; Autonomic Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asymptomatic Individuals (Active Comparator): Individuals aged between 18-50 who volunteered to participate in the study, will form the control group.
  Interventions: Other: VAGUS-NDT
- Individuals with neck pain (Experimental): Individuals with neck pain aged between 18-50 who volunteered to participate in the study, will form the study group.
  Interventions: Other: VAGUS-NDT

INTERVENTIONS:
Other: VAGUS-NDT — Neurodynamic test for vagus nerve

SUMMARY:
The increase in the tension of the soft tissues around a nerve restricts the movement, affects the function of the nerve, and makes the nerve vulnerable to entrapment. Even a mild nerve compression can cause entrapment and lead to neuroinflammation. It is known that inflammatory mediators amplify axonal sensitivity. Although the spontaneous discharge potential of visceral afferents is quite low under normal conditions, neuroinflammation increases the excitability of these fibers. With this mechanism, hyperalgesia may develop in sensory fibers in neuroinflammation. This may cause pathologies in the organs innervated by the relevant nerve.

The fascia and muscles of the cervical region surround the vagus nerve. There are two main fascial compartments in the cervical region. The SCM and trapezius muscle fascias join to the most superficial fascia of the deep cervical fascia and they together form these compartments. These fasciae superiorly attach to the cranium and inferiorly to the pectoral region. The vagus nerve emerges from the jugular foramen together with the 9th and 11th cranial nerves. It then continues through the carotid sheath in the cervical region. The carotid sheath is in contact with the SCM muscle. For this reason, it can be thought that SCM muscle tension or thickness may affect the carotid sheath and thus the function of the vagus nerve passing through it.

In summary, deterioration in vagus nerve activity plays a role in pathologies of the organs innervated by the vagus. Although the relationship between vagal dysfunction and gastrointestinal system symptoms is clear, the mechanisms affecting vagus nerve function have not yet been clarified. It has been reported in the literature that some maneuvers from the cervical region are also effective on the vagus nerve. Also, according to investigators' clinical experience, gastrointestinal symptoms are frequently observed in patients with increased cervical soft tissue tension. However, there are not enough studies investigating whether the cervical region soft tissue tension can affect the gastrointestinal system via the vagus nerve. Therefore, this study was planned to examine the relationship of cervical soft tissue tension with vagus nerve function and gastrointestinal symptoms in asymptomatic individuals and individuals with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Being 18-50 of age,
* Having less than 30 body mass index,
* Being a volunteer

Exclusion Criteria:

* Having any type of malign disease,
* Being diagnosed with a systemic disease (cardiologic, gastrointestinal, rheumatological, neurological, etc.),
* Having any type of surgery within the last 6 months,
* Being diagnosed with Whiplash syndrome
* Having an unhealed fracture
* Pregnancy
* Using prescribed medicine for the gastrointestinal system

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of Vagal Function | 10 minutes, in one assessment session
  Vagus nerve function will be evaluated with the Vagus Neurodynamic Test (VAGUS-NDT). Carta et al. VAGUS-NDT, which was validated and reliable in 2020, evaluates vagal function selectively. The test is performed with the patient in the supine position. The test is considered positive if unpleasant sensations are described when pressure is applied to the abdomen after the head is placed in cervicocranial flexion, lateral flexion, and rotation.
Evaluation of SCM Muscle Tension | 10 minutes, in one assessment session.
  SCM muscle tension will be performed with Myoton-3 (Muomeetria AS, Tallinn, Estonia) myometer. Myometer is a high validity and reliability method used to evaluate muscle tension. During the measurement, the device will give the tension of the muscle numerically by making a light touch on the skin. For the measurement, the myotone will be placed perpendicular to the midpoint between the anterior surface of the manubrium sterni and the mastoid process of the temporal bone, and an average of 10 measurements will be used.
Hospital Anxiety and Depression Scale | 10 minutes, in one assessment session
  Hospital Anxiety and Depression Scale was developed by Zigmond and Snaith, and the Turkish version of the scale was published by Aydemir et al. The scale consists of 14 items, 7 of which assess anxiety and 7 of which assess depression symptoms. It is a 4-point Likert scale type and is scored between 0-3. A high score indicates high levels of anxiety and depression

SECONDARY OUTCOMES:
Evaluation of Neck Disability | 5 minutes, in one assessment session.
  The level of neck disability will be evaluated using the The Neck Disability Questionnaire. It was developed by Vernon et al. as a neck version of the Oswestry Low Back Pain Scale. Within the scope of this study, the Neck Disability Questionnaire will be applied to the participants with a neck pain severity of 3 and above on the Numerical Pain Rating Scale. The Neck Disability Questionnaire includes ten questions about pain, personal care, concentration, work, driving, and sleeping. Each question is scored between 0-5 points. The total score is evaluated out of 50. A high score means a high disability.
Evaluation of Pain Intensity | 1 minutes, in one assessment session.
  Pain intensity will be assessed using the Numerical Pain Rating Scale. The 11-item version of the scale, which is frequently used to measure the severity of pain in adults, will be used. Within the scope of this study, a scale will be used to measure the severity of neck pain of the participants. With this scale, participants will be asked to measure their neck pain on a scale of 0-10. A value of '0' indicates no pain and a value of '10' indicates excruciating pain.
Evaluation of Gastrointestinal Symptoms | 5 minutes, in one assessment session.
  Gastrointestinal symptoms will be evaluated using the Gastrointestinal Symptoms Rating Scale. Revicki et al. The scale developed by CBS measures common symptoms in CBS diseases. A seven-point Likert-type scale consisting of 15 items consisting of five sub-dimensions was made in order. These sub-dimensions are; reflux, indigestion, diarrhea, constipation and abdominal pain. The total score ranges from 15 to 105, with a high score indicating severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Utku Berberoğlu, MSc, Study Chair — Hacettepe University; Özgün Uysal, MSc, Study Chair — Hacettepe University; Özlem Ülger, Professor, Study Director — Hacettepe University
Locations (1):
- Yasemin Özel Aslıyüce, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No